CLINICAL TRIAL: NCT06793956
Title: Open-Label, Phase Ib Study of Sintilimab and Linperlisib Combination Treatment in Patients with Relapsed or Refractory Extranodal Natural Killer/T Cell Lymphoma (NKTCL)
Brief Title: Sintilimab and Linperlisib Combination Treatment in Relapsed or Refractory Extranodal Natural Killer/T Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-753
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Extranodal Natural Killer/T Cell Lymphoma
Keywords: Sintilimab; Linperlisib; Extranodal Natural Killer/T Cell Lymphoma
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab and Linperlisib Combination Treatment (Experimental)
  Interventions: Drug: Sintilimab and Linperlisib Combination Treatment

INTERVENTIONS:
Drug: Sintilimab and Linperlisib Combination Treatment — Sintilimab administered via intravenous infusion; Linperlisib administered orally.

SUMMARY:
This is an open-label, phase Ib study evaluating the combination treatment of sintilimab and linperlisib in patients with relapsed or refractory extranodal natural killer/T-cell lymphoma (NKTCL).

ELIGIBILITY:
Key Inclusion Criteria:

1. Pathologically confirmed extranodal NKTCL.
2. Voluntary participation in the clinical study; fully understand the study, and have signed the written informed consent form.
3. Age ≥ 18 years.
4. Relapsed or refractory NKTCL after failure of at least one line of asparaginase-based chemotherapy or chemoradiotherapy regimen.
5. ECOG performance status: 0-2.
6. Estimated survival time ≥ 3 months.
7. At least one measurable lesion according to the Lugano 2014 lymphoma evaluation criteria.
8. Adequate organ and bone marrow function.

Key Exclusion Criteria:

1. Patients previously treated with PI3K inhibitors.
2. Patients with hemophagocytic syndrome.
3. Patients known to be allergic to any component of monoclonal antibodies.
4. Patients with a history of other malignancies within the past 5 years or concurrent malignancies (excluding basal cell carcinoma of the skin).
5. Patients with aggressive NK-cell leukemia or central nervous system involvement.
6. Patients who have participated in other drug clinical trials within 4 weeks prior to the start of this study or have received anti-tumor treatment within 4 weeks before the study initiation.
7. Patients with clinically significant gastrointestinal abnormalities that may affect drug intake, transport, or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction) or patients who have undergone total gastrectomy.
8. Patients with a history of interstitial lung disease (except for asymptomatic interstitial lung disease caused by radiotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
DLT | Cycle 1 (21 days)
  Dose-limiting toxicity
RP2D | Cycle 1 (21 days)
  Phase II Recommended Dose

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 weeks
  To investigate the antitumor efficacy
AE and SAE | Up to 24 weeks
  Number of participants with adverse events (AE) and severe adverse events (SAE)
2-year Progression-free survival(PFS) | Defined as the proportion of patients without disease progresion, treatment discontinuation, or death for any reason within 24 months of enrollment
  To investigate the antitumor efficacy
2-year Overall survival(OS) | Defined as the proportion of patients without disease progresion, treatment discontinuation, or death for any reason within 24 months of enrollment
  To investigate the antitumor efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided